CLINICAL TRIAL: NCT01249885
Title: Observational Study - Pacifier Use in Israeli Children
Brief Title: Implications of Pacifier Use in Israeli Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Hadas Katz-Sagi, DMD, Hadassah Medical Center
Other Study IDs: 112010hmo-ctil
Record Dates: First submitted 2010-11-28; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Crossbite; Openbite; Drooling
Keywords: pacifier sucking; children; occlusion; drooling
MeSH Terms: conditions — Malocclusion; Open Bite; Sialorrhea; Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to examine pacifier sucking habits among children, and to assess implications of the oral habit - for example malocclusions and drooling. The effect of pacifier sucking will be recorded and compared to pacifier type and frequency of use.

DETAILED DESCRIPTION:
Pacifier study protocol

* The study will take place in children day care centers in Jerusalem and "HaSharon" area.
* First step = Receiving an approval from the Children's parents and the day care management for the research.
* Next step = Examine a total of 400 children who use a pacifier, with a dental mirror in regular lighting condition.
* The procedure is short, no need of repetition or tracing and without any side effects or discomfort.

Part 1- a short questionnaire of demographic background- will be answered by the parents:

1. Personal details- Parents names and ages, child's name and ID number, relation to the child (mother, father…)
2. Social economic status - mother's education, place of residence, number of children in the family.
3. Child's personal details -gender, age, number of siblings
4. Pacifier use habits- period of use, type of pacifier, frequency of use, reason of using a pacifier.
5. Child's Dental condition- drooling, cross bite, open bite.
6. Parents' Awareness of pacifier's effect on mouth development.
7. Parents' approval for child examination. Part 2- clinical- visual examination for identification of relevant findings

1. Child's pacifier type. 2. Dental clinical examination performed in a lightened room:

* Diagnosis of caries- data will be written in a chart.
* Diagnosis of malocclusion- open bite or cross bite 3. Diagnosis of drooling from mouth corners which indicates malocclusion. Redness or dryness around lips and chin can imply drooling.

ELIGIBILITY:
Inclusion Criteria:

* healthy children aged 3-4 years that use a pacifier

Exclusion Criteria:

children suffering from a chronic or developmental disease that can affect the orofacial region

* finger sucking children children suffering from low muscle tonus, abnormal drooling

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 400 children
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated); Study Completion 2013-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Katz-Sagi, DMD, Principal Investigator — Hadassah MO; Diana Ram, DMD, Study Director — Hadassah MO
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel